CLINICAL TRIAL: NCT00926718
Title: The Effect of Rocuronium on the Response of CVI to Laryngoscopy
Brief Title: The Effect of Rocuronium on the Response of Composite Variability Index (CVI) to Laryngoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Vincent's Medical Center (Unknown)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Donald Mathews, MD, Associate Chair, Anesthesiology, Saint Vincents Catholic Medical Centers
Organization: St Vincent's Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: SVCMC_09_021
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Laryngoscopy
Keywords: BIS monitor; rocuronium; The effect of the neuromuscular blocking drug rocuronium on the response of the Composite Variability Index to laryngoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose 1a (Experimental)
  Interventions: Drug: remifentanil infusion
- Dose 2a (Experimental)
  Interventions: Drug: rocuronium dose + remifentanil infusion
- Dose 3a (Experimental)
  Interventions: Drug: rocuronium dose + remifentanil infusion
- Dose 1b (Experimental)
  Interventions: Drug: remifentanil infusion
- Dose 2b (Experimental)
  Interventions: Drug: rocuronium dose + remifentanil infusion
- Dose 3b (Experimental)
  Interventions: Drug: rocuronium dose + remifentanil infusion

INTERVENTIONS:
Drug: remifentanil infusion — rocuronium dose 0 mg/kg + remifentanil infusion of 2ng ml-1
  Arms: Dose 1a
Drug: rocuronium dose + remifentanil infusion — rocuronium dose 0.4 mg/kg+ remifentanil infusion of 2ng ml-1
  Arms: Dose 2a
Drug: rocuronium dose + remifentanil infusion — rocuronium dose 0.6 mg/kg+ remifentanil infusion of 2ng ml-1
  Arms: Dose 3a
Drug: remifentanil infusion — rocuronium dose 0 mg/kg + remifentanil infusion of 8ng ml-1
  Arms: Dose 1b
Drug: rocuronium dose + remifentanil infusion — rocuronium dose 0.4 mg/kg+ remifentanil infusion of 8ng ml-1
  Arms: Dose 2b
Drug: rocuronium dose + remifentanil infusion — rocuronium dose 0.6 mg/kg+ remifentanil infusion of 8ng ml-1
  Arms: Dose 3b

SUMMARY:
Eighty subjects will be recruited from those scheduled for surgery requiring general anesthesia at St Vincent's Hospital. Subjects must have American Society of Anesthesiologists (ASA) status of 1 or 2 (be fairly healthy), a BMI between 18-35 (reasonably healthy weight), and be between the ages of 18 and 75. They will not be eligible if they take certain medications or are expected to have a difficult intubation.

Subjects will be randomized (assigned by chance) to one of four rocuronium doses of 0, 0.2, 0.4, or 0.6 mg kg-1. All are acceptable clinical doses for performing a laryngoscopy. In the operating room, routine monitors will be applied, including a Bispectral Index (BIS) sensor and an M-Entropy sensor. Subjects will receive 0.025 mg kg-1 midazolam (a standard pre-op dose) and will be put to sleep. Once asleep, the subject will receive a rocuronium dose, followed by laryngoscopy three minutes later. The anesthesiologist performing the laryngoscopy will not know what dose of rocuronium the subject received. CVI, entropy, amount of muscle relaxation, and vital signs will be monitored and recorded throughout the procedure.

Subjects will receive propofol and remifentanil infusions during the case. These are commonly used medications for anesthesia. The subjects will also be randomized to two additional groups. One group will receive a remifentanil infusion of 2ng ml-1 and the other group will receive a 8ng ml-1 remifentanil infusion. Both doses are acceptable and often used during standard clinical care. The propofol infusion will be adjusted to keep the BIS number between 45-60. The anesthesiologist will not be able to see the CVI value. The times of certain intraoperative events, such as intubation and incision, will be recorded. All subjects will receive a morphine bolus (0.10-0.15 mg/kg) towards the end to reduce post-operative pain, as per standard clinical care. As the subject wakes up, time to eye opening and orientation will be recorded. The subject will rate their pain on a numerical pain scale and the quality of emergence will be assessed.

Upon arrival in the post anesthesia care unit (PACU), subjects will be asked to rate their pain again using the same pain scale. The pain score will be evaluated every 10 minutes for half an hour, then every hour until they are discharged from PACU.

DETAILED DESCRIPTION:
The Composite Variability Index (CVI, Aspect Medical System, Norwood MA) is a new parameter (measurement) that provides information about the amount of painful stimulation during surgery. It is part of the Bispectral Index (BIS, Aspect Medical Systems, Norwood MA), a well-established and widely used parameter that shows how awake/asleep patients are during general anesthesia and may indicate a need for more medication. The CVI component provides specific information about whether the patient needs pain medication (called opioids) and not just medication that makes you sleep (called hypnotics). The CVI is made of the BIS number and a measure of facial muscle movement (EMG). Both these components increase with painful stimulation, and decrease when pain medication is given.

Neuromuscular blocking drugs (NMD) are paralyzing medications that are often used during surgery to relax the body and make it easier for the surgeon to perform the surgery and the anesthesiologist to insert the breathing tube (called intubation). Facial muscles are resistant to NMD effects, but they might affect the EMG reading, making the CVI less useful when a patient needs NMD. The M-entropy monitor (GE Healthcare, Helsinki, Finland) is similar to the BIS monitor with CVI and is affected by large NMD doses. The purpose of this study is to examine the effect of rocuronium, a NMD, on the response of CVI and M-entropy to laryngoscopy under anesthesia. A laryngoscopy is the standard way of examining and opening the patient's airway before inserting the breathing tube. It is fairly stimulating so anesthesiologists sometimes, but not always, administer a NMD (in varying doses) before performing the laryngoscopy in standard care.

Eighty subjects will be recruited from those scheduled for surgery requiring general anesthesia at St Vincent's Hospital. Subjects must have ASA status of 1 or 2 (be fairly healthy), a BMI between 18-35 (reasonably healthy weight), and be between the ages of 18 and 75. They will not be eligible if they take certain medications or are expected to have a difficult intubation.

Subjects will be randomized (assigned by chance) to one of four rocuronium doses of 0, 0.2, 0.4, or 0.6 mg kg-1. All are acceptable clinical doses for performing a laryngoscopy. In the operating room, routine monitors will be applied, including a BIS sensor and an M-Entropy sensor. Subjects will receive 0.025 mg kg-1 midazolam (a standard pre-op dose) and will be put to sleep. Once asleep, the subject will receive a rocuronium dose, followed by laryngoscopy three minutes later. The anesthesiologist performing the laryngoscopy will not know what dose of rocuronium the subject received. CVI, entropy, amount of muscle relaxation, and vital signs will be monitored and recorded throughout the procedure.

Subjects will receive propofol and remifentanil infusions during the case. These are commonly used medications for anesthesia. The subjects will also be randomized (assigned by chance) to two additional groups. One group will receive a remifentanil infusion of 2ng ml-1 and the other group will receive a 8ng ml-1 remifentanil infusion. Both doses are acceptable and often used during standard clinical care. The propofol infusion will be adjusted to keep the BIS number between 45-60. The anesthesiologist will not be able to see the CVI value. The times of certain intraoperative events, such as intubation and incision, will be recorded. All subjects will receive a morphine bolus (0.10-0.15 mg/kg) towards the end to reduce post-operative pain, as per standard clinical care. As the subject wakes up, time to eye opening and orientation will be recorded. The subject will rate their pain on a numerical pain scale and the quality of emergence will be assessed.

Upon arrival in the PACU, subjects will be asked to rate their pain again using the same pain scale. The pain score will be evaluated every 10 minutes for half an hour, then every hour until they are discharged from PACU. The total dose of pain medications administered in PACU will be recorded. Upon PACU discharge, subjects will be asked to rate their overall experience with anesthesia. Demographic data will also be collected. All data will be kept in locked file cabinets and study results will be shared with research personnel at Aspect Medical Systems.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ASA physical status class I or II. (This will exclude subjects with significant medical problems).
* Body mass index between 18 and 35 kg m-2.
* No use of psychotropic or neuropsychiatric medications.
* A airway assessment with no indication of a difficult intubation including a class I or II Malampatti airway and a mandible-to-hyoid distance of greater than three fingerbreadths.
* Age between 18-75 years.

Exclusion Criteria:

* Does not meet inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Variable response to medication given. | 1-6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Vincent Catholic Medical Centers, New York, New York, United States